CLINICAL TRIAL: NCT06888050
Title: Efficacy and Safety of Henagliflozin Proline and Metformin Hydrochloride Extended-release Tablets (Ⅰ) Versus Metformin Tablets in Patients With New-onset Type 2 Diabetes: a Multicenter, Randomized Controlled Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Collaborators: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KT20240056
Record Dates: First submitted 2025-03-10; First posted 2025-03-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-03

CONDITIONS: New-onset Type 2 Diabetes
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- henagliflozin proline and metformin hydrochloride extended-release tablets (Ⅰ) (Experimental): Start with henagliflozin proline and metformin hydrochloride extended-release tablets (Ⅰ) (5mg/500mg, once a day, two tablets at a time) + raw live-style intervention
  Interventions: Drug: henagliflozin proline and metformin hydrochloride extended-release tablets (Ⅰ)
- metformin (Active Comparator): Initiation of metformin (500 mg twice a day) + lifestyle intervention
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: henagliflozin proline and metformin hydrochloride extended-release tablets (Ⅰ) — henagliflozin proline and metformin hydrochloride extended-release tablets (Ⅰ) (5mg/500mg, once a day, two tablets each time) plus lifestyle intervention
  Arms: henagliflozin proline and metformin hydrochloride extended-release tablets (Ⅰ)
Drug: Metformin — Metformin (500mg, twice a day) plus lifestyle intervention
  Arms: metformin

SUMMARY:
This multicenter, randomized controlled trial aims to evaluate the efficacy and safety of Henagliflozin-Metformin Sustained-Release Tablets (I) versus Metformin Tablets in newly diagnosed type 2 diabetes mellitus (T2DM). A total of 268 participants will be randomized (1:1) into two groups: the experimental group receiving Henagliflozin-Metformin Sustained-Release Tablets (I) (5mg/500mg, once daily) with lifestyle intervention, and the control group receiving Metformin Tablets (500mg, twice daily) with lifestyle intervention. The primary outcome is the change in glycated hemoglobin (HbA1c) from baseline at 24 weeks. Secondary outcomes include changes in fasting/postprandial blood glucose, body weight, metabolic parameters, diabetes remission rate, and safety assessments. This trial will provide evidence for early combination therapy in newly diagnosed T2DM patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years old.
* Diagnosed with type 2 diabetes according to WHO diagnostic criteria, with HbA1c between 7% and 9% at this examination, fasting venous blood glucose ≤ 11.1 mmol/L, and BMI ≥ 18.5 kg/m2; known disease duration ≤ 24 months.
* Voluntary participation in this study and signing of the informed consent form. If the subject is unable to read the informed consent form (e.g., illiterate subjects), a witness must be present to observe the informed consent process and sign the informed consent form on their behalf.
* No previous use of hypoglycemic drugs.

Exclusion Criteria:

* Type 1 diabetes.
* Participants who have participated in other clinical trials of diabetes treatment drugs before the start of this study.
* Those who have experienced diabetic ketoacidosis, diabetic lactic acidosis or hyperosmolar non-ketotic coma within the past six months and required hospitalization.
* Those who have experienced decompensated heart failure (NYHA class III and IV), unstable angina, stroke or transient ischemic attack, myocardial infarction, severe arrhythmia, undergone cardiac surgery or vascular reconstruction (including coronary artery bypass grafting or percutaneous coronary intervention) within the past six months.
* Those taking glucocorticoid drugs (excluding topical or inhaled medications).
* Those with a life expectancy of less than one year due to malignant tumors, active tuberculosis, or acute infections.
* Those with clinically significant urinary tract or genital infections, or a history of recurrent urinary tract or genital infections.
* Those with a history of hypertension whose blood pressure has not been effectively controlled despite antihypertensive drug treatment: systolic blood pressure (SBP) > 160 mmHg and/or diastolic blood pressure (DBP) > 100 mmHg.
* Those with liver and kidney function indicators meeting the following criteria: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥ 3.0×ULN; estimated glomerular filtration rate (eGFR) < 45 ml/min/1.73 m² (calculated according to the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula).
* Those allergic to the investigational drug or its components.
* Pregnant or lactating women and those with the intention to conceive within three months of the last dose.
* Other patients deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Glycosylated Hemoglobin, Type A1C（HbA1C） | 24 weeks

SECONDARY OUTCOMES:
Fasting blood glucose (FBG) | 4,12, 24 weeks
2-hour postprandial blood glucose (PBG) | 4,12, 24 weeks
Diabetes reversal rate | 36 weeks
fasting insulin/C-peptide and postprandial 2-hour insulin/C-peptide | 24 weeks
HbA1c | 4, 12weeks
Blood lipids (high-density lipoprotein cholesterol [HDL-C], low-density lipoprotein cholesterol [LDL-C], triglycerides [TG]) | 12, 24 weeks
blood urine acid | 12, 24 weeks
Urinary Albumin-to-Creatinine Ratio (UACR) | 12, 24 weeks
body weight | 4,12, 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No